CLINICAL TRIAL: NCT02609412
Title: Immediate Effects of Self-myofascial Release on Latent Trigger Point Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Dr. Winfried Banzer, Head of Department, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SpM2015-002
Record Dates: First submitted 2015-10-02; First posted 2015-11-20 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Trigger Points

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Static compression of LMTRP (Experimental): static compression of most sensitive LMTRP with the foam roll for 90 seconds
  Interventions: Other: Static compression of LMTRP
- Dynamic self-myofascial release of calf (Experimental): dynamic self-myofascial release rolling back and forth on the entire calf for 90 seconds with the foam roll
  Interventions: Other: Dynamic self-myofascial release of calf
- Placebo laser acupuncture of LMTRP (Placebo Comparator): placebo laser acupuncture applied on most sensitive LMTRP of the calf, light and acoustic sounds provided, but laser remains switched off, 90 seconds
  Interventions: Device: Placebo laser acupuncture of LMTRP

INTERVENTIONS:
Other: Static compression of LMTRP — Static compression of most sensitive Triggerpoint with a foam roller (Blackroll Inc., Germany).
  Arms: Static compression of LMTRP
Other: Dynamic self-myofascial release of calf — Dynamic self-massage of the calf with a foam roller (Blackroll Inc., Germany).
  Arms: Dynamic self-myofascial release of calf
Device: Placebo laser acupuncture of LMTRP — Used device: Laserneedle System (Laserneedle Systems GmbH, Glienicke/Nordbahn, Germany). Electrodes positioned on skin but device remains switched off.
  Arms: Placebo laser acupuncture of LMTRP

SUMMARY:
Latent myofascial trigger points (LMTRP) which impair neuromuscular performance occur in both, patients and asymptomatic subjects. As evidence suggests that LMTRP can transform into active trigger points, therapy seems warranted. Besides other modalities, self-massage using foam rollers (self-myofascial release) has been applied as a treatment. However, there is no data on the efficacy of this method concerning LMTRP. Thus, the present study aims to evaluate the effects of different forms of self-myofascial release on LMTRP pain.

Healthy patients with LMTRP in the calf are randomly allocated to one of three groups: 1) 90s static compression of the most sensitive LMTRP by means of the foam roll, 2) dynamic self-myofascial release rolling back and forth on the calf muscles for 90s using a foam roller, 3) placebo laser acupuncture of the most sensitive LMTRP. All subjects participate in a familiarization session with the foam roller one week prior to treatments. As an outcome, pressure pain threshold is assessed with an algometer. The investigators hypothesize, that static compression can reduce pressure pain of LMTRP more effective than dynamic self-myofascial release. The investigators further expect that placebo treatment will be the least effective method.

ELIGIBILITY:
Inclusion Criteria:

* at least one diagnosed latent myofascial trigger point in the calf
* age 18 to 65 years
* written informed consent

Exclusion Criteria:

* active myofascial trigger point in the calf
* regular intake of drugs or within past 48 hours
* severe psychiatric, neurological, orthopaedic, cardiovascular or endocrine diseases
* pregnancy or nursing period
* any condition that negatively influences current quality of life

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in pressure pain threshold [kg/cm²] assessed by pressure algometer | Baseline (M1) - 3 minutes (M2)

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Banzer, MD, PhD, Principal Investigator — Department of Sports Medicine, Goethe University Frankfurt/Main
Locations (1):
- Goethe University Frankfurt/Main, Frankfurt am Main, Germany